CLINICAL TRIAL: NCT03682445
Title: Metabolic, Physical Responses To Exercise In Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, GULIN FINDIKOGLU, Associate Professor, MD, PhD, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GFindikoglu
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Type2 Diabetes Mellitus; Exercise
Keywords: Type 2 diabetes mellitus; exercise; aerobic; interval; continuous
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study has 3 arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants wil be making exercise. It is not possible to make participants blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity interval exercise (Active Comparator): Participants with type 2 Diabetes mellitus in High intensity interval exercise (HIIE) group will make aerobic exercise using bicycle at high intensity followed by low intensity periods under observation in the hospital.
  Interventions: Other: exercise
- Moderate intensity continuous exercise (Active Comparator): Participants with type 2 Diabetes mellitus in Moderate intensity continuous exercise (MIC) group will make aerobic exercise using bicycle at moderate intensity during the session under observation in the hospital.
  Interventions: Other: exercise
- Control group (No Intervention): The participants in the control group will make stretching exercise at home

INTERVENTIONS:
Other: exercise — Aerobic tyep of exercise will be made at different intensities in 2 groups.
  Arms: High intensity interval exercise; Moderate intensity continuous exercise

SUMMARY:
The aim of this study is to compare the effects of high intensity interval exercise and moderate intensity continuous exercise on metabolic parameters, physical measures, fitness level, body composition and miRNA-143 level in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Volunteers with type 2 diabetes mellitus will be evaluated in terms of any contra-indication that will restrain them from making exercise. 90 male or female volunteers who are suitable in terms of inclusion/exclusion criteria will be invited for the study. Volunteers will be randomly distributed to one of the 3 groups. Each group will contain 30 participants. 1. group will make aerobic exercise which is in the form of high intensity interval exercise 2.group will make aerobic exercise which is in the form of moderate intensity continuous exercise 3. Control group. Exercise groups will be cycling under observation in the hospital setting. Control group will make simple stretching exercises at home. Participants will be requested to complete a 3 months of exercise. They will be evaluated before and at the end of the 3 months of exercise with physical measures such as waist and hip circumference, fitness level measured by exercise testing, body composition measured by bioimpedance, metabolic parameters such as blood glucose level, HbA1C and measured by blood tests.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have type 2 Diabetes mellitus less than 10 years and more than 1 year.
2. Participants must have appropriate medical therapy and diet.
3. Participants must not be treated with insulin.
4. Participants must be exercising less than 210 minutes/ week.

Exclusion Criteria:

1. Participants with prominent cardiovascular disease
2. Participants with coronary artery disease
3. Participants with moderate to severe valvular disease
4. Participants with atrial fibrillation
5. Participants with untreated hypertension
6. Participants with congenital heart disease
7. Participants with retinopathy
8. Participants with neuropathy
9. Participants with macro albuminuria
10. Participants with cerebrovascular disease
11. Participants with ejection fraction less than 40
12. Participants with body mass index greater than 35.
13. Participants with prominent ischemic changes in EKG at rest or during exercise.
14. Participants with cigarette or alcohol addiction
15. Participants on drugs that interferes with body fat distribution (such as insulin, thiazolidinediones)

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c level. | 12 weeks
  Change in HbA1c level measured in the blood after exercise compared to beginning

CONTACTS AND LOCATIONS:
Overall Officials: Gulin Findikoglu, Assoc Prof, Principal Investigator — pamukkale university, Medical Faculty, PMR Department
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Findikoglu G, Altinkapak A, Yaylali GF. Is isoenergetic high-intensity interval exercise superior to moderate-intensity continuous exercise for cardiometabolic risk factors in individuals with type 2 diabetes mellitus? A single-blinded randomized controlled study. Eur J Sport Sci. 2023 Oct;23(10):2086-2097. doi: 10.1080/17461391.2023.2167238. Epub 2023 Feb 5. PMID 36622777